CLINICAL TRIAL: NCT03515603
Title: Compare Between Endoscopic and Microsurgical Transsphenoidal Resection of Pituitary Adenomas With Intraoperative MRI
Brief Title: Endocrine Outcome of Surgery for Pituitary Adenoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruiting
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Andrej Pala, Principal Investigator, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EndOSPA
Record Dates: First submitted 2018-04-14; First posted 2018-05-03 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Intervention Model Description: prospective randomized
Who Masked: Participant, Care Provider
Masking Description: only surgeon knows the used technique, endocrinologist, patient and all involved medical staff is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- microsurgical technique (Active Comparator)
  Interventions: Procedure: Microsurgical resection
- endoscopic technique (Active Comparator)
  Interventions: Procedure: Endoscopic resection

INTERVENTIONS:
Procedure: Endoscopic resection — Transsphenoidal endoscopic resection of pituitary adenoma
  Arms: endoscopic technique
Procedure: Microsurgical resection — Transsphenoidal microsurgical resection of pituitary adenoma
  Arms: microsurgical technique

SUMMARY:
Prospective and randomized compare between microsurgical and endoscopic transsphenoidal MRI assisted resection of pituitary adenomas.

DETAILED DESCRIPTION:
The main aim of the study is to compare microsurgical and endoscopic transsphenoidal surgery and to determine endocrine outcome. Secondary extent of resection and quality of life will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Suspected symptomatic or progressively growing pituitary adenoma
* Informed consent

Exclusion Criteria:

* Prolactinoma
* No follow-up possible
* Emergency surgery without informed consent or without intraoperative MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
endocrine function | 1 year after surgery
  Testing of pituitary function with insulin-hypoglycemic test, results will be dichotomized as satisfactory or not satisfactory. Satisfactory outcome is defined, if pituitary function improves or is stable, if compared to preoperative testing.

SECONDARY OUTCOMES:
Extent of resection | tumor volume before the surgery, 3 months after surgery
  Volumetric analysis of tumor volume before the surgery, intraoperatively and 3 months after surgery will be performed. Gross total resection is defined as no tumor present in gadolinium enhanced T1 sequences
Quality of Life, EQ-5D | 3 months and 1 year after surgery
  EQ-5D will be evaluated before surgery, after the surgery in 3 months and after 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Pala, MD, Principal Investigator — University Ulm, Department of Neurosurgery
Locations (1):
- Department of Neurosurgery, Günzburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pala A, Grubel N, Mayer B, Becker R, Sommer F, Schmitz B, Etzrodt-Walter G, Wirtz CR, Hlavac M. Endocrine Outcome and Quality of Life After Transsphenoidal Resection of Pituitary Adenoma-A Prospective Randomized Single-Blinded Study Comparing Endoscopic Versus Microscopic Resection. Neurol Int. 2025 Jan 10;17(1):5. doi: 10.3390/neurolint17010005. PMID 39852769